CLINICAL TRIAL: NCT04020926
Title: Impact of Hyponatremia on Muscle Strength, Gait and Balance, and Cognitive Function: a Prospective Observational Study
Brief Title: Impact of Hyponatremia on Muscle Strength, Gait and Cognitive Function
Status: Terminated | Type: Observational
Why Stopped: Study was stopped due to COVID-19 pandemic.
Sponsor: Bürgerspital Solothurn (Other)
Responsible Party: Principal Investigator, LINDNER Gregor, Director Dept. of Internal and Emergency Medicine, Bürgerspital Solothurn
Other Study IDs: 2019-00650
Record Dates: First submitted 2019-07-10; First posted 2019-07-16 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Hyponatremia
Keywords: hyponatremia
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study patients with hyponatremia, defined as a serum sodium < 126 mmol/L on admission to the hospital will be tested for muscular power by use of a hand grip dynamometer, for cognitive function by use of the Montreal-Cognitive-Assessment and gait stability by use of the Tinetti test. The tests will be performed on admission as well es after correction of hyponatremia.

DETAILED DESCRIPTION:
The investigators broad objective is to examine in a prospective study whether an association exists between hyponatremia and psychomotor deficits. The specific aims are:

A.) To measure muscle strength by use of a dynamometer in patients presenting with moderate to severe hyponatremia (serum sodium ≤ 125 mmol/L) at the emergency department before and after correction of hyponatremia (serum sodium ≥ 135 mmol/L).

B.) To test for balance and gait disorders before and after correction of hyponatremia C.) To investigate whether presence of hyponatremia is associated with cognitive impairment that isreversible after correction of serum sodium.

The hypothesis is that hyponatremia is associated with reduced muscle strength, impaired balance, and cognitive impairment, and that the correction of the serum sodium will lead to an improvement of these parameters.

Design & Setting

The investigators will conduct a single-center, prospective, observational study at the General Hospital Solothurn. The study will be conducted at the Department of Emergency Medicine, where patients will be screened for hyponatremia, and the Department of General Internal Medicine, where screening will occur both in the inpatient and outpatient services.

If a serum sodium of 125 mmol/L is detected in a blood sample sent from the Department of Emergency Medicine or General Internal Medicine, the Center for Laboratory Medicine will notify the study team responsible for patient enrollment using a dedicated pager. Then, a member of the study team will approach potential participants, inform them about the study goals and procedures, obtain informed consent, and enroll them into the study. Patients enrolled in the Department of Emergency Medicine needing hospitalization will primarily hospitalized in the Department of General Internal Medicine, unless hospitalization at specialist ward is indicated.

Patient enrollment criteria

Inclusion criteria Consecutive patients aged 18 years or above presenting with moderately to severe hyponatremia (serum sodium ≤ 125 mmol/L after correction for blood glucose), who give informed consent.

Exclusion criteria

* Patients who do not give or are not able to give informed consent.
* Patients with concomitant Potassium dysregulation (K+<3.5 mmol/l or K+>5.0 mmol/l)

Baseline data collection

1. Clinical data Of all patients included in the study, data on age, sex, comorbidities, and current medications taken by the patients will be gathered.
2. Serum sodium measurements Measurements of serum sodium will be performed through the Center for Laboratory Medicine of the General Hospital Solothurn. Sodium determination will be performed by use of ion-selective electrode using the ICT (Na+, K+, Cl-) Sample Diluent Kit, Abbott Laboratories, Chicago, IL, USA. Additionally, serum osmolality, potassium, magnesium, calcium, creatinine, albumin and hemoglobin will be measured. All of these parameters are standard measurements in case of a severe electrolyte disorder and are part of clinical practice in the care for patients with electrolyte disorders. All laboratory parameters will be measured at baseline and after correction of serum sodium. In order to avoid multiple blood drawings for the patient the parameters mentioned above will be reordered from blood already taken for serum sodium determination.

Endpoints A.) Muscle strength in pounds and kilogram before and after correction of hyponatremia.

B.) Results for the Tinetti performance-oriented mobility assessment (POMA) to evaluate static and dynamic balance abilities during and after correction of hyponatremia.

C.) Results for the Montreal Cognitive Assessment (MOCA) test to assess mild cognitive impairment before and after correction of hyponatremia.

Muscle strength at handgrip will be measured at time of presentation at the clinic with a serum sodium ≤ 125 mmol/L and 24 to 48 hours after correction of hyponatremia at a serum sodium ≥ 135 mmol/L using the Jamar ® hydraulic hand dynamometer, Lafayette Instrument, Lafayette, IN, USA. Strength will be measured in pounds and kilograms thrice at baseline and after correction of hyponatremia, respectively. The best result of each test will be used for the analysis. The test will be conducted by either Drs. Woitok or Lindner.

The Tinetti POMA, a simple, easily administered test, will be used to measure patients' gait and balance taking about 10 to 15 minutes. Scoring of the Tinetti Assessment Tool is done on a three point ordinal scale with a range of 0 to 2. A score of 0 represents the most severe impairment, while a 2 would represent patient independence. The individual scores are then combined to form three measures; an overall gait assessment score, an overall balance assessment score, and a gait and balance score. The test has been validated in several studies and found to be a useful screening tool for gait instabilities and prediction of falls. The Tinetti POMA form is shown in the Appendix. The test will be performed at baseline and 24 to 48 hours after correction of hyponatremia. The test will be conducted by the study team.

The MOCA is a 30-point test administered in about 10 minutes designed to identify mild cognitive impairment. The test is validated for a large variety of diseases ranging from frontotemporal dementia to HIV or chronic obstructive pulmonary disease. The MOCA form is shown in the Appendix. The test will be performed at baseline and 24 to 48 hours after correction of hyponatremia. The test will be conducted by the study team.

Correction of hyponatremia Correction of hyponatremia will be performed at the discretion of the attending physician depending on the etiology of hyponatremia. Hypovolemic hyponatremia (diuretic induced hyponatremia, gastrointestinal fluid losses, low solute intake) will be corrected by use of an isotonic crystalloid to replenish volume deficits and in a next step, if needed, by use of loop diuretics to increase free water excretion and simultaneous substitution of fluid losses by isotonic crystalloids until normonatremia (i.e. serum sodium ≥ 135 mmol/L) is reached. If hyponatremia is due to adrenal insufficiency steroids will be applied in addition to volume resuscitation by use of isotonic crystalloids. In case of the syndrome of inappropriate anti diuretic hormone secretion water restriction will be ordered initially. Hyponatremia due to low effective circulating volume (heart failure, cirrhosis of the liver) will be corrected by salt and water restriction. Serum sodium corrections will be accompanied by frequent monitoring of serum sodium concentration. The study team will provide the managing physician at the ward current expert recommendations on the correction of hyponatremia in order to ensure best treatment for all study patients.

Sample size Sample size was calculated on basis of the MOCA test. To achieve a power of 90% and a two-sided alpha level of 0.05, the sample size needed to detect a difference of 5 points (shown difference between normal individuals and those with mild cognitive impairment) between the baseline and post-correction MOCA scores would be 44 patients. Thus, we plan to enroll a total of 50 patients.

Statistical analysis Data will be presented as means and standard deviation or medians and interquartile range as appropriate. Wilcoxon signed ranked tests will be used to compare results on muscle strength, Tinetti score and MOCA scores, since those are not normally distributed and samples will be dependent since every patient serves as his own control. A p-value of ≤ 0.05 will be considered statistically significant. Statistics will be calculated using SPSS Statistics, IBM Inc., Armonk, NY, USA.

Study period Based on general Patient count and prevalence of Hyponatremia, the enrollment of the sample size of 50 patients seems realistic in a 12-month period, starting on 01 September 2019.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or above
* serum sodium ≤ 125 mmol/L
* informed consent.

Exclusion Criteria:

* age < 18 years
* not give or are not able to give informed consent
* K+<3.5 mmol/l
* K+>5.0 mmol/l)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: We will include all consecutive patients >/= 18 years with a serum sodium level < 126 mmol/L on admission to the Hospital who give consent.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Muscle strength | Correction of hyponatremia (up to 1 week).
  A.) Change in muscle strength in kilogram before and after correction of hyponatremia.
Mobility assessment | Correction of hyponatremia (up to 1 week).
  B.) Change in results for the Tinetti performance-oriented mobility assessment (POMA) to evaluate static and dynamic balance abilities during and after correction of hyponatremia.
Cognitive Function | Correction of hyponatremia (up to 1 week).
  C.) Change in results for the Montreal Cognitive Assessment (MOCA) test to assess mild cognitive impairment before and after correction of hyponatremia.

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Lindner, M.D., Principal Investigator — Dept. of Internal and Emergency Medicine, Buergerspital Solothurn, Switzerland
Locations (1):
- Buergerspital Solothurn, Solothurn, Canton of Solothurn, Switzerland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT04020926/Prot_000.pdf